CLINICAL TRIAL: NCT07277881
Title: The Effect of Reversal of Remimazolam Sedation With Flumazenil on Cognitive Function in Patients Undergoing Hip Arthroplasty Under Spinal Anesthesia
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Principal Investigator, Cezary Kapłan, resident, Medical University of Gdansk
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 429/2025
Record Dates: First submitted 2025-11-16; First posted 2025-12-11 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Delirium; Sedation; Remimazolam; Hip Arthroplasty, Total
MeSH Terms: conditions — Emergence Delirium | interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Flumazenil Group (Experimental): Patients will receive a single intravenous bolus of 0.5 mg of flumazenil
  Interventions: Drug: remimazolam sedation reversal with flumazenil
- Placebo Group (Placebo Comparator): Patients will receive a single intravenous bolus of 0.9% NaCl
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: remimazolam sedation reversal with flumazenil — Immediately after the skin suture is completed, before leaving the operating room, the patient will receive an intravenous bolus administered over 30 seconds containing the contents of a pre-prepared, coded syringe with flumazenil
  Arms: Flumazenil Group
Drug: placebo — Immediately after the skin suture is completed, before leaving the operating room, the patient will receive an intravenous bolus administered over 30 seconds containing the contents of a pre-prepared, coded syringe with placebo (0,9% NaCl)
  Arms: Placebo Group

SUMMARY:
This clinical trial aims to establish whether reversing remimazolam sedation with flumazenil can prevent postoperative neurocognitive disorders in patients undergoing total hip replacement surgery. The main questions it aims to answer are:

* Does administering flumazenil after surgery lead to an improvement in cognitive function (measured by the MoCA scale) at 24 hours post-operation compared to a placebo?
* Does this intervention reduce the incidence of postoperative delirium within the first 48 hours? Researchers will compare flumazenil to a placebo (0.9% saline solution) to see if actively reversing sedation leads to better cognitive outcomes and a lower incidence of delirium.

Participants will:

* Undergo a planned total hip replacement surgery under spinal anesthesia.
* Receive sedation with remimazolam during the operation.
* At the end of the surgery, receive an intravenous injection of the study drug (flumazenil) or a placebo.
* Undergo assessments for cognitive function (using the MoCA scale) and delirium (using the 4AT scale) before and at multiple time points after the surgery.
* Complete a questionnaire about their quality of recovery (QoR-15).

ELIGIBILITY:
Inclusion Criteria:

* Patient qualified for elective, primary, unilateral, total hip replacement.
* Patient assessed on the ASA I-III scale.
* MoCA score obtained during screening ≥ 23 points (to exclude patients with significant pre-existing cognitive impairment).
* Ability to understand information about the study and express informed, written consent to participate.

Exclusion Criteria:

* Known hypersensitivity or allergy to benzodiazepines, flumazenil, local anesthetics
* Contraindications to spinal anesthesia or patient refusal of this anesthesia technique.
* Severe liver dysfunction.
* History of epilepsy or seizures
* Chronic (daily use for > 2 weeks in the last 3 months) use of benzodiazepines or non-benzodiazepine hypnotics (so-called "Z" drugs: zolpidem, zopiclone, zaleplon).
* Alcohol abuse defined as regular consumption of more than: in men: 40 g of pure ethanol at a time; in women: 20 g of pure ethanol at a time, or a history of psychoactive substance dependence.
* Planned revision hip arthroplasty or bilateral surgery.
* Significant neurological or psychiatric diseases that may affect the assessment of cognitive function.
* The need for sedative premedication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | from baseline (preoperative) to 24 hours after surgery
  The MoCA is a cognitive screening tool. The total score ranges from 0 to 30 points. A higher score indicates better cognitive function.

SECONDARY OUTCOMES:
Incidence of delirium (defined as a score of ≥ 4 on the 4AT scale) | within the first 48 hours after surgery, assessed every 6 hours.
Total duration of delirium episodes in hours | within the first 48 hours after surgery
Preoperative Anxiety Level assessed by Amsterdam Preoperative Anxiety and Information Scale (APAIS) | baseline (preoperative)
  The Amsterdam Preoperative Anxiety and Information Scale (APAIS) is a questionnaire consisting of 6 items graded on a 5-point Likert scale (ranging from 1 = "not at all" to 5 = "extremely"). The total score ranges from 6 to 30. A higher score indicates higher levels of preoperative anxiety.
Montreal Cognitive Assessment (MoCA) score | at 1 and 6 hours after surgery
  The MoCA is a cognitive screening tool. The total score ranges from 0 to 30 points. A higher score indicates better cognitive function.
Mini Montreal Cognitive Assessment (mini-MoCA) scores (telephone assessment) | at 3 and 6 months after surgery
  mini-MoCA is an abbreviated version of the MoCA used for remote assessment. The total score usually ranges from 0 to 15 points. A higher score indicates better cognitive function.
Quality of Recovery-15 (QoR-15) Questionnaire Score | at 24 hours after surgery
  The QoR-15 is a patient-reported outcome measure assessing the quality of recovery after anesthesia and surgery. The total score ranges from 0 to 150. A higher score indicates a better quality of recovery.
The duration of hospital stay | Assessed up to 30 days post-surgery (or through hospital discharge, whichever occurs first).
  measured in days from the date of surgery to the date of hospital discharge.
Maximum and average pain intensity measured by Numeric Rating Scale (NRS) at the following time points | 6, 12, 24, and 48 hours after surgery
  Pain intensity will be assessed using the Numeric Rating Scale (NRS). The scale ranges from 0 to 10, where 0 indicates "no pain" and 10 indicates "worst pain imaginable".
Total oxycodone consumption (in mg) | during the first 48 hours after surgery
Mean bispectral index (BIS) during sedation and percentage of time within the optimal range (60-80) | during surgery
Total dose of remimazolam administered (in mg) | during surgery
Dose of vasopressor drugs | during surgery
Need for additional sedative drugs | during surgery